CLINICAL TRIAL: NCT07364825
Title: Behavioral Health Home Hospital: A Pilot Randomized Controlled Trial
Brief Title: Acute Psychiatric Care at Home for Lower-risk Patients With Acute Psychiatric Illness Who Require Inpatient Care
Acronym: BHH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: The Thompson Family Foundation Inc (Unknown)
Responsible Party: Principal Investigator, David Levine, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P001301
Record Dates: First submitted 2026-01-07; First posted 2026-01-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Psychosis; Anxiety; Depression; Behavioral and Psychiatric Symptoms of Dementia
Keywords: behavioral health home hospital; home hospital; hospital in the home; hospital at home
MeSH Terms: conditions — Psychotic Disorders; Anxiety Disorders; Depression; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral health home hospital Care (Experimental): Patients receive hospital level psychiatric care in their home
  Interventions: Other: Behavioral Health Home Hospital

INTERVENTIONS:
Other: Behavioral Health Home Hospital — Patients receive hospital level psychiatric care in their home

SUMMARY:
The goal of this pilot randomized controlled trial is to learn if adult patients with acute psychiatric conditions can receive hospital-level care at home. The main question it aims to answer is:

What percentage of eligible patients agree to enroll and be randomized to behavioral health home hospital (intervention) or the brick-and-mortar hospital (control)?

DETAILED DESCRIPTION:
Behavioral Health Home Hospital (BHH) aims to investigate the feasibility of providing acute psychiatric care at home for a highly selected lower-risk subset. Eligible patients will be admitted to behavioral health home hospital. Subjects include a highly selected lower-risk subset of patients (18 years of age or older) that require hospitalization for an acute psychiatric condition, caregivers (18 years of age or older) of the highly selected lower-risk subset of patients that require hospitalization of an acute psychiatric condition, and clinicians that provide care to intervention and control patients.

ELIGIBILITY:
General patient inclusion criteria:

≥18 years old

Resides or will reside during hospital care within a 10-mile geographic area surrounding BWFH or BWH.

Patients must be able to be safely managed at home with the in-home clinical coverage and monitoring provided by the BHH program, as determined by the BHH MD. If the BHH MD determines that caregiver support is required for safe participation, the patient must have a caregiver who is able to provide the required level of support to be eligible for enrollment. The level of caregiver support will be determined on a case-by-case basis by the patient's clinical team and BHH MD based on the patient's clinical presentation, safety needs, and functional status (see section 6.1 for details)

To participate in the study, the patient must agree to the level of in-home support and monitoring determined by the study doctor and clinical team. This could include the possibility of asking the patient to agree to be in the same home with their caregiver 24/7 during their entire hospitalization.

Patient clinical inclusion criteria

Voluntarily consent to BHH admission (patient or proxy consent; if proxy consents, patient assents)

Requires hospital-level care for anxiety/depression, psychosis, or behavioral and psychological symptoms of dementia (BPSD)

No current restraint use

No catatonia

Has capacity to consent OR can assent to study and has proxy who can consent Does not need in person socialization that cannot be provided remotely

Can reliably communicate with the BHH team (self or caregiver)

Does not need safety monitoring more frequently than every 30 minutes

Medical condition(s) manageable by BHH

Is not a risk of harm to others, and meets the following criteria:

Has not harmed staff in the past

Consider excluding for a score >1 on the Broset Violence Checklist

Consider prior harm to others; determine context surrounding prior harm, consider other collateral information from family, friends, and other providers

Is not a risk of harm to self, and meets the following criteria:

SAFE-T Protocol with a Columbia-Suicide Severity Rating Scale (C-SSRS) that is low or moderate risk

No evidence of alcohol intoxication or risk of severe withdrawal

No active substance use or if substance use then they can abstain during hospitalization (Consider any active treatment plan, type of substance used, and access to substances)

Consider previous suicide attempts, intensity, lethality, and compulsivity of self-harm behaviors when determining eligibility

Patient does not have behaviors that would prevent them from being cared for at home:

Modified Agitation Severity Scale (MASS) score < 6

Does not have lack of insight or severe disorganization

Pittsburgh Agitation Scale score < 3. Consider excluding the patient for a score of 3 or 4.

Patient diagnosis-specific inclusion criteria:

If patient has a diagnosis of psychosis:

They have NOT developed ideas/beliefs which are significantly detached from the shared beliefs of others

If patient has a diagnosis of BPSD, patient must:

Have an identifiable treatment goal Be willing and able to participate in therapeutic care Agree to wear the Angelsense device

Patient environmental inclusion criteria:

HITS Screening Tool for Domestic Violence (requires patient interview) negative

Is not in police custody

Is not undomiciled

Does not reside in a skilled nursing facility, long term acute care hospital, or detoxification facility

Residence has the capacity to be therapeutic and has working heat (Oct-Apr), working air conditioner if forecast >80 F (Jun-Sep), running water, electricity, and no suspected bed bugs, lice, or scabies

No direct access to a firearm (even if stored)

No illicit drugs in the home

Willing and able to secure pets during BHH visits

Willing to secure medications and other substances, including marijuana, in a BHH lockbox during BHH

Has access to their home (e.g., keys to get into their house)

Caregiver inclusion criteria (caregiver is not required to participate in the study; if a caregiver does enroll in the study, the following inclusion criteria apply)

Age >= 18 years old

Has capacity to consent to study

Clinician inclusion criteria

A BHH clinical team member (a clinician providing care in the home, in-person or remotely).

Or a clinician at the hospital providing care to a control patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Patient randomization | Date of patient admission, expected one day
  Total number and % of eligible patients who agree to enroll and be randomized

SECONDARY OUTCOMES:
Caregivers' perceptions and attitudes towards being a caregiver assessed through semi-structured interviews with caregivers | Date of discharge to 30 days post discharge, assessed up to 2 months
  Secondary
Clinicians' perceptions and attitudes towards providing care to their patients through semi-structured interviews with caregivers | Date of enrollment to date of final discharge, assessed up to 4 months
  Secondary
Percent of patients that recommend their hospital stay | Day of discharge to 30 days after discharge, assessed up to 2 months
  Secondary
Patients' perceptions and attitudes towards their hospitalization | Date of discharge to 30 date after discharge, assessed up to 2 months
  Semi-structured interview with patients (control & intervention patients) to assess subjects' perceptions and attitudes towards their hospitalization
Caregiver refusal rate and reasons for refusal | Date of patient admission, expected one day
  Secondary
Patient refusal rate and reasons for refusal | Date of patient admission, expected one day
  Secondary
Perceived clinician acceptability | Date of enrollment to date of final discharge, assessed up to 4 months
  Mean or median score of clinician recommend care score (scale from 0-10)
Perceived patient acceptability | Date of discharge, an expected average of 7 days after the date of admission
  Mean or median score of patient recommend care score (scale from 0-10)
Total number of caregivers screened | On the date of patient recruitment, expected one day
  Total number of caregivers screened through caregiver screening forms completed
Patient's C-SSRS low or moderate risk (yes/no) | On the date of patient recruitment, expected one day
  Secondary
Patient not reside in a skilled nursing facility, long term acute care hospital, or detoxification facility (yes/no) | On the date of patient recruitment, expected one day
  Secondary
Patient not in police custody (yes/no) | On the date of patient recruitment, expected one day
  Secondary
Patient not undomiciled (yes/no) | On the date of patient recruitment, expected one day
  Secondary
Patient not ≦19 weeks pregnant AND does not need fetal monitoring / not pregnant (yes/no) | On the date of patient recruitment, expected one day
  Secondary
Patient not catatonic (yes/no) | On the date of patient recruitment, expected one day
  Secondary
Patient does not require restraints (yes/no) | On the date of patient recruitment, expected one day
  Secondary
Patient reside in the catchment area (yes/no) | On the date of patient recruitment, expected one day
  Secondary
Patient employment status | On the date of patient recruitment, expected one day
  Secondary
Patient race/ethnicity | On the date of patient recruitment, expected one day
  Secondary
Patient sex assigned at birth | On the date of patient recruitment, expected one day
  Secondary
Patient Age | On the date of patient recruitment, expected one day
  Secondary
Patient diagnosis | On the date of patient recruitment, expected one day
  Secondary
Reasons for patient ineligibility | On the date of patient recruitment, expected one day
  Reasons for ineligibility, %
Reasons for caregiver ineligibility | On date of recruitment, expected one day
  Reasons for ineligibility, %
Total number and % of patients consented to study | On date of enrollment, expected one day
  Secondary
Total number and % of caregivers consented to study | On date of enrollment, expected one day
  Secondary
Percentage of patient consent forms completed properly | On date of enrollment, expected one day
  Consent forms with the patient name and signature, the consenting clinician signature, and date and time
Percentage of caregiver verbal consent completed properly | On the date of enrollment, expected one day
  Documentation that verbal consent was completed appropriately, signature of the person obtaining consent, and date and time of the verbal consent
Randomization procedures followed for each patient | On the date of admission, expected one day
  Consent form complete before randomization and the patient receiving the treatment they were allocated to
Total number and % of patients withdrew from the study | From date of admission to date of discharge, an expected average of 7 days
  Secondary
Total number and % of patients who complete hospitalization | From date of admission to date of discharge, an expected average of 7 days
  Secondary
Total number and % of caregivers who withdrew from the study | From date of admission to date of discharge, an expected average of 7 days
  Secondary
Total number and % of caregivers who stayed with the patient through entire hospitalization | From date of admission to date of discharge, an expected average of 7 days
  Intervention arm only
Total number and % of patients lost to follow-up | Day of discharge to 30 days later
  Secondary
Total number and % of caregivers lost to follow up | Day of discharge to 30 days later
  Secondary
% of patients that received intended intervention | From date of admission to date of discharge, an expected average of 7 days
  2 visits per day by RN, 1 daily visit by physician
% of patients that received 2 RN visits per day | From date of admission to date of discharge, an expected average of 7 days
  Secondary
% of patients who received one daily remote visit by a physician | From date of admission to date of discharge, an expected average of 7 days
  Secondary
% of patients in possession of prohibited contraband | From date of admission to date of discharge, an expected average of 7 days
  Secondary
% of patients who received intended number of mental health checks | From date of admission to date of discharge, an expected average of 7 days
  Secondary
% of questions missed in admission, discharge, and post-discharge surveys | At admission, at discharge (expected average of 7 days after admission), and at 30 days after discharge
  Secondary
% of patients who complete all surveys | At admission, at discharge (expected average of 7 days after admission), and at 30 days after discharge
  Secondary
% of questions missed in caregiver admission and discharge surveys | At admission and at discharge (expected average of 7 days after admission)
  Secondary
% of caregivers who complete all surveys | At admission, at discharge (expected average of 7 days after admission), and at 30 days after discharge
  Secondary
% of patients, caregivers, and clinicians who complete interviews | Date of enrollment to date of final discharge, assessed up to 4 months
  Secondary
% of missing data | At admission, at discharge (expected average of 7 days after admission), and at 30 days after discharge
  % of patients missing EHR data, cost data, activity data or Redcap data
Total number of patients assessed for eligibility | On the date of patient recruitment, expected one day
  Total number and % of patients initially screened that were approached and not approached.
Total number of caregivers assessed for eligibility | On the date of patient recruitment, expected one day
  Total number and % of caregivers initially screened that were approached and not approached
Eligible patients approached and not approached | On the date of recruitment, expected one day
  Total number and % of patients approached and not approached that met all eligibility criteria for the study
Eligible caregivers approached and not approached | On the date of patient recruitment, expected one day
  Total number and % of caregivers approached and not approached that met all eligibility criteria for the study

OTHER OUTCOMES:
Time between patient being approached by RA and consent signature | Date of enrollment, expected one day
  Operational Process Measures
Total direct cost | Day of patient admission to 30 days post discharge
  Total direct cost, direct cost of the acute care episode, direct cost of post-discharge period and direct cost post-randomization.
Length of stay | Date of admission to date of discharge, expected average of 7 days
  Measured by the days in the brick and mortar compared to in-home days and the total length of stay
Length of stay, date and time | Date of admission to date of discharge, expected average of 7 days
  Date and time presented to the ED and admitted to the hospital (brick-and-mortar or behavioral health home hospital
Length of stay, early transfer | Date of admission to date of discharge, expected average of 7 days
  For intervention arm only, date and time that the patient left the brick-and-mortar and date and time that the patient arrived home
EuroQol-5D-5L and Euro-VAS change in score | At admission, at discharge (the day the patient leaves the hospital environment, expected average of 7 days after admission), and at 30 days after discharge
  Change in score at 30 days compared with enrollment
EuroQol-5D-5L and Euro-VAS percent improvement in each milestone | At admission, at discharge (the day the patient leaves the hospital environment, expected average of 7 days after admission), and at 30 days after discharge
  Measured compared to the minimal important difference (at least 0.037 index for the EuroQol-5D-5L
Number of mental health specialist checks per day | From date of admission to date of discharge, an expected average of 7 days
  Acute episode utilization
Ratio of observed versus expected mental health specialist checks | From date of admission to date of discharge, an expected average of 7 days
  Acute episode utilization
Percent utilized social work | From date of admission to date of discharge, an expected average of 7 days
  Acute episode utilization
Percent utilized consultant | From date of admission to date of discharge, an expected average of 7 days
  Acute episode utilization
Percent utilized urgent mobile integrated health visits | From date of admission to date of discharge, an expected average of 7 days
  Acute episode utilization
Percent utilized virtual group therapy | From date of admission to date of discharge, an expected average of 7 days
  Acute episode utilization
Percent utilized 1:1 virtual therapy | From date of admission to date of discharge, an expected average of 7 days
  Acute episode utilization
Total number of patients screened | On the date of patient recruitment, expected one day
  Total number of patients screened through number of patient screening forms completed
Percent utilized virtual reality group therapy | From date of admission to date of discharge, an expected average of 7 days
  Acute episode utilization
Average number of enrollments per day | At the end of the study, assessed up to 2 months
  Operational Process Measures
Percent utilized 1:1 virtual reality therapy | From date of admission to date of discharge, an expected average of 7 days
  Acute episode utilization
Percent utilized virtual reality therapeutic activities | From date of admission to date of discharge, an expected average of 7 days
  Acute episode utilization
Time to readmission, days | Day of discharge to 30 days later
  Post discharge 30-day utilization
Percent readmission to inpatient psychiatry | Day of discharge to 30 days later
  Post discharge 30-day utilization
Percent readmission to hospital for non-psychiatric illness | Day of discharge to 30 days later
  Post discharge 30-day utilization
Percent emergency department visit | Day of discharge to 30 days later
  Post discharge 30-day utilization
Percent observation stay | Day of discharge to 30 days later
  Post discharge 30-day utilization
Percent outpatient psych visits | Day of discharge to 30 days later
  Post discharge 30-day utilization
Percent primary care provider visits | Day of discharge to 30 days later
  Post discharge 30-day utilization
Calories per day | Date of admission to date of discharge, expected average of 7 days
  Exploratory
Percent wear time of the Actigraph | Date of admission to date of discharge, expected average of 7 days
  Exploratory
Percent sleep per day | Date of admission to date of discharge, expected average of 7 days
  Exploratory
Percent time low physical activity | Date of admission to date of discharge, expected average of 7 days
  Exploratory
Percent time moderate-vigorous physical activity | Date of admission to date of discharge, expected average of 7 days
  Exploratory
Percent time walking | Date of admission to date of discharge, expected average of 7 days
  Exploratory
Percent time sedentary | Date of admission to date of discharge, expected average of 7 days
  Exploratory
Number of steps | Date of admission to date of discharge, expected average of 7 days
  Exploratory
Percent top-box response to Picker survey questions | Date of discharge, assessed up to 2 months
  Exploratory
Mean Global experience (scale 0-10 about the patient's hospital experience) | Date of discharge, assessed up to 2 months
  Exploratory
Mean patient recommend care | Date of discharge, assessed up to 2 months
  Exploratory
Mean net promoter score (% of those who recommend minus the % of those who don't recommend) | Date of discharge, assessed up to 2 months
  Exploratory
Percent patients with any adverse events | Date of patient admission to date of patient discharge, expected average of 7 days
  Exploratory
Percent of patients with psychiatry-related adverse events | Date of patient admission to date of patient discharge, expected average of 7 days
  Exploratory
Percent of patients with non-psychiatry-related adverse events | Date of patient admission to date of patient discharge, expected average of 7 days
  Exploratory
Percent intervention patients transferred back to hospital for adverse events | Date of patient admission to date of patient discharge, expected average of 7 days
  Intervention patients that were admitted to the BAM because of their adverse event and their number of days in BAM
Percent of intervention patients round trip from BAM to behavioral health home hospital | Date of patient admission to date of patient discharge, expected average of 7 days
  Due to a safety event but transferred back home to complete their BHH admission and number of days in BAM
Number of days spent entirely at home | Day of discharge to 30 days later
  Exploratory
Caregiver burden overall score | Date of admission to date of discharge, an expected average of 7 days
  Assessed through the Zarit Burden Interview - short form where >13 points is considered the cut-off score
Percent of providers reporting burnout | Date of enrollment to date of final discharge, assessed up to 4 months
  Measured through the Mini-Z survey and a score of 3 or higher on the question about burnout
Time between admission to BHH and arrival home (intervention) or transfer to ward (control) | At patient enrollment, expected average of one day
  Operational Process Measures
Average transport time | Date of admission to date of discharge, an expected average of 7 days
  Operational Process Measures
Caregiver burden percent moderate-to-severe or severe burden | Date of admission to date of discharge, an expected average of 7 days
  Assessed through the Zarit Burden Interview - short form where >13 points is considered the cut-off score
Time between arriving home to evaluation by nurse (intervention only) | On date of admission, expected average of one day
  Operational Process Measures
Minutes per day spent in 1:1 virtual therapy | Date of admission to date of discharge, expected average of 7 days
  Exploratory
Minutes per day spent in virtual group therapy | Date of admission to date of discharge, expected average of 7 days
  Exploratory
Minutes per day spent in 1:1 virtual reality therapy | Date of admission to date of discharge, expected average of 7 days
  Exploratory
Minutes per day spent in virtual reality group therapy | Date of admission to date of discharge, expected average of 7 days
  Exploratory
Minutes per day spent in virtual reality activities | Date of admission to date of discharge, expected average of 7 days
  Exploratory
Average time of visit (non-admission and non-discharge) | Date of admission to date of discharge, expected average of 7 days
  Operational Process Measures
Gender | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Primary language | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Health insurance status, public/private/none | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
BMI | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Comorbidities, type and # | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Partner status | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Education | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
9-digit zip code | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Smoking status | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Medications used as outpatient, number | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
DNR/I code status | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Lives alone | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Admission source | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Admitting Diagnosis | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Number of non-psychiatric admissions in the previous 6 months | Date of admission, assessed up to 2 months]
  Patient Co-variates of Interest
Number of psychiatric admissions in the previous 6 months | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Number of psychiatric ED visits in the previous 6 months | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Number of non-psychiatric ED visits in the previous 6 months | Date of admission, assessed up to 2 months
  Patient co-variate of interest
Primary care provider | Date of admission, assessed up to 2 months
  Patient co-variate of interest
Home health aide prior to admission | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
BRIEF health literacy screening tool | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Taking psychiatric medication, yes/no | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Length of psychiatric condition, years | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Alcohol use by average drinks per week | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Substance use disorder yes/no | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Type of substance use disorder (OUD, AUD, CUD, other) | Date of admission, assessed up to 2 months
  Patient Co-variates of Interest
Length of diagnosis, years | Date of admission, assessed up to 2 months
  Co-variates for patients diagnoses
Type of anxiety, psychosis, depressive or BPSD diagnosis | Date of admission, assessed up to 2 months
  Co-variates for patients
Anxiety severity for people with diagnosis of anxiety | At admission, at discharge (expected average of 7 days after admission), and at 30 days after discharge
  Measured through the generalized anxiety disorder-7 item
Psychosis severity | At admission, at discharge (expected average of 7 days after admission), and at 30 days after discharge
  Measured through the BPRS
History of suicide | Day of admission, assessed up to 2 months
  Co-variate for Patients with Depression
Suicidal ideation (based off C-SSRS) | Day of admission, assessed up to 2 months
  Co-variates for Patients with Depression
Depression severity, PHQ-9 score | At admission, at discharge (expected average of 7 days after admission), and at 30 days after discharge
  Co-variates for Patients with Depression
BPSD severity, quick dementia rating system (QDRS) | Day of admission, assessed up to 2 months
  Co-variates for Patients with BPSD
Frail scale | Day of admission, assessed up to 2 months
  Co-variates for Patients with BPSD
Clinician age | Day of admission, assessed up to 2 months
  Clinician Co-variates of Interest
Clinician role | Day of admission, assessed up to 2 months
  Clinician Co-variates of Interest
Clinician number of years in practice | Day of admission, assessed up to 2 months
  Clinician Co-variates of Interest
Clinician gender | Day of admission, assessed up to 2 months
  Clinician Co-variates of Interest
Clinician race | Day of admission, assessed up to 2 months
  Clinician Co-variates of Interest
Clinician ethnicity | Day of admission, assessed up to 2 months
  Clinician Co-variates of Interest
Caregiver Age | Day of admission, assessed up to 2 months
  Caregiver Co-variates of Interest
Caregiver relationship to the patient | Day of admission, assessed up to 2 months
  Caregiver Co-variates of Interest
Primary caregiver yes/no | Day of admission, assessed up to 2 months
  Caregiver Co-variates of Interest
Paid caregiver yes/no | Day of admission, assessed up to 2 months
  Caregiver Co-variates of Interest
Caregiver employment status | Day of admission, assessed up to 2 months
  Caregiver Co-variates of Interest
Caregiver lives with patient | Day of admission, assessed up to 2 months
  Caregiver Co-variates of Interest
Caregiver education | Day of admission, assessed up to 2 months
  Caregiver Co-variates of Interest
Caregiver race | Day of admission, assessed up to 2 months
  Caregiver Co-variates of Interest
Caregiver ethnicity | Day of admission, assessed up to 2 months
  Caregiver Co-variates of Interest
Caregiver partner status | Day of admission, assessed up to 2 months
  Caregiver Co-variates of Interest
Capacity to consent (yes/no) | Date of recruitment, expected average one day
  Caregiver Co-variates of Interest
Agree to stay with the patient 24/7 while they are hospitalized to provide support (yes/no) | Date of recruitment, expected average one day
  Caregiver Co-variates of Interest
Willing to respond and help the patient in an urgent need (yes/no) | Date of recruitment, expected average one day
  Caregiver Co-variates of Interest
Concerns about safety or interpersonal/environmental triggers for the patient (yes/no) | Date of recruitment, expected average one day
  Caregiver Co-variates of Interest
Caregiver will need help in areas (yes/no) | Date of recruitment, expected average one day
  Caregiver Co-variates of Interest
Caregiver has medications and/or substances to secure during BHH (yes/no) | Date of recruitment, expected average one day
  Caregiver Co-variates of Interest
Caregiver feels physically and emotionally prepared to provide caregiver services (yes/no) | Date of recruitment, expected average one day
  Caregiver Co-variates of Interest
Caregiver meets eligibility (yes/no) | Date of recruitment, expected average one day
  Caregiver Co-variates of Interest
Reasons for ineligibility (if ineligible) | Date of recruitment, expected average one day
  Caregiver Co-variates of Interest
Wants to participate in the research surveys and interview (yes/no) | Date of recruitment, expected average one day
  Caregiver Co-variates of Interest

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - McLean Hospital, Belmont, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Jamaica Plain, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levine DM, Ouchi K, Blanchfield B, Saenz A, Burke K, Paz M, Diamond K, Pu CT, Schnipper JL. Hospital-Level Care at Home for Acutely Ill Adults: A Randomized Controlled Trial. Ann Intern Med. 2020 Jan 21;172(2):77-85. doi: 10.7326/M19-0600. Epub 2019 Dec 17. PMID 31842232